CLINICAL TRIAL: NCT02296801
Title: A Phase II Randomized Study Evaluating the Biological and Clinical Effects of the Combination of Palbociclib With Letrozole as Neoadjuvant Therapy in Post-Menopausal Women With Estrogen-Receptor Positive Primary Breast Cancer
Acronym: PALLET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Pfizer (Industry); Royal Marsden NHS Foundation Trust (Other); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-11; WI180455 (Other: Pfizer)
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Breast Carcinoma; Breast Tumors
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A: letrozole (Active Comparator): letrozole 2.5 mg tablet orally daily for 14 weeks
  Interventions: Drug: Letrozole
- B: letrozole then letrozole + palbociclib (Experimental): letrozole 2.5 mg orally daily plus beginning 2 weeks after starting letrozole, palbociclib 125 mg capsule orally daily for 1 week then 1 week off, then a 3 weeks on and 1 week off cycle for a total of 14 weeks from start of letrozole therapy
  Interventions: Drug: Letrozole; Drug: palbociclib
- C: palbociclib then letrozole + palbociclib (Experimental): palbociclib 125 mg capsule orally daily (for a 3 weeks on and 1 week off cycle for a total of 14 weeks from start of palbociclib) plus beginning 2 weeks after starting palbociclib, letrozole 2.5 mg tablet orally daily for a total of 12 weeks from start of letrozole therapy
  Interventions: Drug: Letrozole; Drug: palbociclib
- D: letrozole + palbociclib (Experimental): letrozole 2.5 mg tablet orally daily for a total of 14 weeks plus palbociclib 125 mg capsule orally daily for a 3 weeks on and 1 week off cycle, for a total of 14 weeks from start of therapy
  Interventions: Drug: Letrozole; Drug: palbociclib
- Combined Groups B+D+C (Other): Combined data
  Interventions: Drug: Letrozole; Drug: palbociclib

INTERVENTIONS:
Drug: Letrozole
Drug: palbociclib
  Arms: B: letrozole then letrozole + palbociclib; C: palbociclib then letrozole + palbociclib; Combined Groups B+D+C; D: letrozole + palbociclib

SUMMARY:
This study will look at effects the combination of palbociclib and letrozole may have on estrogen receptor (ER)-positive/human epidermal growth factor receptor 2 (HER2)-negative breast cancer tumors which have not yet been treated. Letrozole is a type of endocrine therapy called an aromatase inhibitor (AI) and is standard treatment for post-menopausal women with ER-positive/HER2-negative breast cancer.

DETAILED DESCRIPTION:
The FB-11 study is a Phase II, randomized, open label, four arm study to examine the biological and clinical effect of neoadjuvant letrozole with or without palbociclib in the first-line treatment of estrogen-receptor (ER) positive, HER2-negative early invasive breast cancer. The co-primary aims of this study are to to compare the changes in the proliferation marker Ki67, and to compare clinical response after 14 weeks of therapy with letrozole with or without palbociclib.

The FB-11 study initiative is a joint partnership between the NSABP Foundation, Inc. (NSABP) Department of Site and Study Management (DSSM) and United Kingdom (UK) co-investigators at the Royal Marsden NHS Foundation Trust and the Institute of Cancer Research (ICR). Parallel protocols will be conducted in the US and Canada (FB-11), and the UK (PALLET) with joint analysis of interim and final data.

Postmenopausal women, newly diagnosed with ER-positive/HER2-negative early breast cancer, who are suitable candidates for neoadjuvant endocrine therapy will be invited to join the FB-11/PALLET trial. Approximately 306 patients will be accrued to this study. Each collaborative group will recruit at least 1/3 and no more than 2/3 of the target accrual.

Patients will be randomized to one of four treatment arms (3:2:2:2 ratio). Treatment in the first 14 weeks of neoadjuvant therapy will be:Arm A Letrozole alone; Arm B Letrozole for 2 weeks followed by letrozole + palbociclib to week 14; Arm C Palbociclib for 2 weeks followed by letrozole + palbociclib to week 14; Arm D Letrozole + palbociclib to week 14.

Letrozole will be administered orally as a 2.5mg daily tablet. Palbociclib will be administered orally as 125mg capsules, daily on a schedule of 3 weeks (21 days) on, 1 week (7 days) off of a 4 week [28 day] cycle.

The end of study therapy for patients in Arm A will be completion of week 14. Patients in Arms B, C, and D will complete study therapy following 14 days of palbociclib in the final treatment cycle past 14 weeks if treatment delays have occurred.

Note: After week 14 (end of study therapy) all patients should continue letrozole until surgery. Letrozole is not considered study therapy beyond completion of week 14 for Arm A or after 14 days of palbociclib in the final treatment cycle for patients in Arms B, C, and D.

Following completion of study therapy, surgery will be scheduled for 15-18 weeks post-randomization. Post-surgical treatment will be at discretion of treating clinician, following local protocols, and not influenced by allocation of treatment within the FB-11/PALLET study.

Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be postmenopausal women defined as: Age 56 or older with no spontaneous menses for at least 12 months prior to study entry; or Age 55 or younger with no menses for at least 12 months prior to study entry (e.g., spontaneous or secondary to hysterectomy) and with a documented estradiol level in the postmenopausal range according to local institutional/laboratory standard; or Age greater than or equal to 18 with documented bilateral oophorectomy.
* Operable ER-positive/HER2- negative, invasive early breast cancer, suitable for neoadjuvant AI treatment. HER2-negative as determined by American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) guidelines.
* No known severe hypersensitivity reactions to compounds similar to palbociclib or palbociclib excipients or to endocrine treatments.
* A breast tumor with an ultrasound size of at least 2.0 cm.
* Patients must have the ability to swallow oral medication.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* At the time of randomization, blood counts performed within 4 weeks prior to randomization must meet the following criteria: absolute neutrophil count (ANC) must be greater than or equal to 1500/mm3; Platelet count must be greater than or equal to 100,000/mm3; Hemoglobin must be greater than or equal to 10 g/dL.
* international normalized ratio (INR) must be within normal limits of the local laboratory ranges.
* The following criteria for evidence of adequate hepatic function performed within 4 weeks prior to study entry must be met: total bilirubin must be less than or equal to upper limit of normal (ULN) for the lab unless the patient has a bilirubin elevation greater than ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and alkaline phosphatase must be must be less than or equal to 1.5 x ULN for the lab; and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be less than or equal to 1.5 x ULN for the lab.
* Serum creatinine performed within 4 weeks prior to study entry must be less than or equal to 1.25 x ULN or estimated creatinine clearance less than 60 mL/min (as calculated using the method standard for the institutions).

Exclusion Criteria:

* Active hepatitis B or hepatitis C with abnormal liver function tests.
* HIV positive patients receiving antivirals.
* Premenopausal or peri-menopausal women.
* Inflammatory/inoperable breast cancer.
* HER2-positive as determined using ASCO-CAP Guidelines.
* Concurrent use (defined as use within 4 weeks prior to baseline tissue sample being taken) of hormone replacement therapy (HRT) or any other estrogen-containing medication (including vaginal estrogens)
* Prior endocrine therapy for breast cancer.
* Any invasive malignancy within previous 5 years (other than basal cell carcinoma or cervical carcinoma in situ).
* Other nonmalignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow up such as: Active infection or chronic infection requiring chronic suppressive antibiotics; Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function; Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids); Seizure disorders requiring medication.
* Diagnosis by fine needle aspiration (FNA) alone or excisional biopsy or lumpectomy performed prior to study entry.
* Surgical axillary staging procedure prior to study procedure (with exception of FNA or core biopsy).
* Definitive clinical or radiologic evidence of metastatic disease.
* History of ipsilateral invasive breast cancer regardless of treatment or ipsilateral ductal carcinoma in situ (DCIS) treated with radiotherapy or contralateral invasive breast cancer at any time.
* Any treatment, including radiotherapy, chemotherapy, and/or targeted therapy, administered for the currently diagnosed breast cancer prior to study entry.
* Use of any medication or substances that are strong inhibitors or inducers of CYP3A isoenzymes.
* Class III or Class IV myocardial disease as described by the New York Heart Association; a recent history (within 6 months) of myocardial infarction, or symptomatic arrhythmia at the time of randomization. Class III: Patients with cardiac disease resulting in marked limitation of physical activity. Such patients are comfortable at rest. Less than ordinary physical activity that causes fatigue, palpitation, dyspnea, or anginal pain. Class IV: Patients with cardiac disease resulting in inability to perform any physical activity without discomfort. Symptoms of cardiac insufficiency or anginal syndrome may be present even at rest.
* QTc greater than 480 msec or a family or personal history of long or short QT syndrome, Brugada syndrome or know history of QTc prolongation, or Torsade de Pointes (TdP).
* The investigator should assess the patient to determine if she has any psychiatric or addictive disorder or other condition that, in the opinion of the investigator, would preclude her from meeting the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2015-01; Primary Completion 2018-07 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (52):
- United States (19):
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - University of Miami Hospital and Clinics - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Norton Healthcare Pavillion, Louisville, Kentucky
  - Norton Cancer Institute - Suburban, Norton Medical Plaza II, Louisville, Kentucky
  - Norton Cancer Institute - Brownsboro Medical Plaza I, Louisville, Kentucky
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Hope Women's Cancer Centers, Asheville, North Carolina
  - Providence Oncology and Hematology Clinic, Portland, Oregon
  - Pinnacle Health Ortenzio Cancer Center, Mechanicsburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Sentara Martha Jefferson Hospital-Phillips Family Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Canada (4):
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - CHU de Quebec - Universite Laval, Québec, Quebec
- United Kingdom (29):
  - Milton Keynes Hospital, Milton Keynes, Buckinghamshire
  - Hinchingbrooke Hospital, Huntingdon, Cambridgeshire
  - Royal Cornwall Hospital, Treliske, Truro, Cornwall
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Royal Sussex County Hospital, Brighton, East Sussex
  - Southend Hospital, Westcliff-on-Sea, Essex
  - Darent Valley Hospital, Dartford, Kent
  - Maidstone Hospital, Maidstone, Kent
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - James Paget University Hospital, Great Yarmouth, Norfolk
  - Musgrove Park Hospital, Taunton, Somerset
  - Weston General Hospital, Weston-super-Mare, Somerset
  - The Royal Marsden Hospital, Sutton, Surrey
  - Salisbury Hospital, Salisbury, Wiltshire
  - Kidderminster Hospital, Kidderminster, Worcestershire
  - Alexandra Hospital, Redditch, Worcestershire
  - Worcestershire Royal Hospital, Worcester, Worcestershire
  - Belfast City Hospital, Belfast
  - Royal Bournemouth Hospital, Bournemouth
  - Western General Hospital (Edinburgh Cancer Centre), Edinburgh
  - St James' University Hospital, Leeds
  - Barnet Hospital, London
  - Whittington Hospital, London
  - University College London Hospitals, London
  - The Royal Marsden Hospital, London
  - Charing Cross Hospital, London
  - Nottingham University Hospitals NHS Trust, City Campus, Nottingham
  - Derriford Hospital, Plymouth
  - Singleton Hospital, Swansea

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Letrozole: letrozole 2.5 mg tablet orally daily for 14 weeks
  Letrozole
- B: Letrozole Then Letrozole + Palbociclib: letrozole 2.5 mg orally daily plus beginning 2 weeks after starting letrozole, palbociclib 125 mg capsule orally daily for 1 week then 1 week off, then a 3 weeks on and 1 week off cycle for a total of 14 weeks from start of letrozole therapy
  Letrozole
  palbociclib
- C: Palbociclib Then Letrozole + Palbociclib: palbociclib 125 mg capsule orally daily (for a 3 weeks on and 1 week off cycle for a total of 14 weeks from start of palbociclib) plus beginning 2 weeks after starting palbociclib, letrozole 2.5 mg tablet orally daily for a total of 12 weeks from start of letrozole therapy
  Letrozole
  palbociclib
- D: Letrozole + Palbociclib: letrozole 2.5 mg tablet orally daily for a total of 14 weeks plus palbociclib 125 mg capsule orally daily for a 3 weeks on and 1 week off cycle, for a total of 14 weeks from start of therapy
  Letrozole
  palbociclib
Period: Overall Study
Arm/Group | A: Letrozole | B: Letrozole Then Letrozole + Palbociclib | C: Palbociclib Then Letrozole + Palbociclib | D: Letrozole + Palbociclib
Started | 103 | 68 | 69 | 67
Completed | 83 | 53 | 50 | 58
Not Completed | 20 | 15 | 19 | 9

BASELINE CHARACTERISTICS:
Population: This population contains all patients who received at least one dose of each of their randomized treatments (i.e. one dose of letrozole for group A, one dose of each of letrozole and palbociclib for groups B.C and D). The as-treated population are used in analyses of assessment of safety and tolerability.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Letrozole | B: Letrozole Then Letrozole + Palbociclib | C: Palbociclib Then Letrozole + Palbociclib | D: Letrozole + Palbociclib | Total
Number analyzed (Participants) | 103 | 68 | 69 | 67 | 307
Age, Customized [Count of Participants; unit: Participants]
  Age 40-49 | 0 | 0 | 1 | 0 | 1
  Age 50-59 | 32 | 15 | 19 | 22 | 88
  Age 60-69 | 34 | 31 | 29 | 30 | 124
  Age 70-79 | 30 | 14 | 17 | 12 | 73
  Greater than or equal to 80 | 7 | 8 | 3 | 3 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 68 | 69 | 67 | 307
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-British-UK patients | 48 | 32 | 28 | 30 | 138
  White-Other-UK patients | 5 | 1 | 7 | 2 | 15
  Indian-UK patients | 0 | 0 | 2 | 1 | 3
  Other Asian background-UK patients | 0 | 2 | 0 | 1 | 3
  Caribbean-UK patients | 1 | 1 | 0 | 1 | 3
  Other Black backgroud-UK patients | 1 | 0 | 0 | 0 | 1
  Other-UK-patients | 1 | 0 | 0 | 0 | 1
  Data not received-UK patients | 0 | 1 | 0 | 1 | 2
  White-Not hispanic/latino-NA patient | 38 | 25 | 26 | 27 | 116
  White-Hispanic/latino-NA patient | 4 | 1 | 1 | 1 | 7
  White-Not known-NA patient | 1 | 0 | 2 | 1 | 4
  Black or African American-NA patient | 1 | 2 | 1 | 0 | 4
  Asian-patient-NA patient | 1 | 1 | 1 | 1 | 4
  Other-patient-NA patient | 1 | 1 | 1 | 0 | 3
  Data not received-NA patient | 1 | 1 | 0 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 47 | 31 | 32 | 31 | 141
  United Kingdom | 56 | 37 | 37 | 36 | 166

OUTCOME MEASURES:

1. Primary Outcome: Measurement of the Proliferation Marker Ki67 (% Positive Tumor Cells)
Description: The change in Ki67 from baseline to 14 weeks.
Time Frame: Baseline and at 14 weeks
Population: Paired Ki67 data from baseline and end of treatment were available for 190 patients. Patients treated with letrozole with palbociclib, i.e. groups B+C+D, were pooled and compared to those treated with letrozole alone (group A). The pooling of groups B-D was pre-planned and defined in the Statistical Analysis Plan.
Measure: Median (Inter-Quartile Range); unit: log fold change in Ki67
Groups:
- B, C + D Palbociclib + Letrozole Regimen: Comparison between Group A and Group (B,C+D).
Arm/Group | A: Letrozole | B, C + D Palbociclib + Letrozole Regimen
Number analyzed (Participants) | 65 | 125
log fold change in Ki67 | -2.2 [-3.4 to -1.0] | -4.1 [-5.0 to -2.8]

2. Primary Outcome: Clinical Response : Number of Patients Who Have Resolution of Measurable Lesions or no New Lesions or Other Signs of Disease Progression Compared to Baseline.
Description: Clinical Response is assessed by ultrasound at the end of the treatment (week 14) according to ECOG response criteria defined in Appendix A1 of the protocol. Number of participants with clinical complete response.
Time Frame: Baseline and at 14 weeks
Population: Clinical response data were available for 279 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | A: Letrozole | B: Letrozole Then Letrozole + Palbociclib | C: Palbociclib Then Letrozole + Palbociclib | D: Letrozole + Palbociclib | B, C + D Palbociclib + Letrozole Regimen
Number analyzed (Participants) | 93 | 63 | 61 | 62 | 186
Participants | 46 | 31 | 35 | 35 | 101

3. Secondary Outcome: Pathological Complete Response (pCR): Number of Patients With no Lesions in Breast and Nodes at Time of Surgery
Description: Pathologic complete response in the breast (pCR breast) is defined as no histologic evidence of invasive tumour cells in the surgical breast specimen. Pathologic complete response in breast and axillary lymph nodes as well as non-axillary SN (pCR breast & nodes) is defined as no histologic evidence of invasive tumour cells in the surgical breast specimen, axillary nodes, or SNs identified after neoadjuvant treatment. Data shows the pCR rates by randomised group.
Time Frame: 14 weeks
Population: There is response data for 279 patients. Patients treated with letrozole with palbociclib, i.e. groups B+C+D, were pooled and compared to those treated with letrozole alone (group A). The pooling of groups B-D was pre-planned and defined in the Statistical Analysis Plan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A: Letrozole | B, C + D Palbociclib + Letrozole Regimen
Number analyzed (Participants) | 91 | 187
percentage of participants | 0.0 [0.0 to 4.0] | 1.1 [0.0 to 3.8]

4. Secondary Outcome: Preoperative Endocrine Prognostic Index (PEPI) Score:
Description: The PEPI score estimates the risk of cancer recurrence after treatment. Analysis of the PEPI score were pre-specified in the protocol and statistical analysis plan. However, pathological/biomarker characteristics which comprise this score such as the Allred score for ER status were not collected during the trial so cannot be calculated at this stage. PEPI Scale range is 0-16 for RFS. Higher score represents worse outcome. No combination of subscales.
Time Frame: 14 weeks
Population: 194 patients have ER, Ki67, tumour size and nodal status available. Patients treated with letrozole with palbociclib, i.e. groups B+C+D, were pooled and compared to those treated with letrozole alone (group A). The pooling of groups B-D was pre-planned and defined in the Statistical Analysis Plan.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- B,C+D Palbociclib +Letrozole Regimen: Comparison between Group A & Group B,C+D
Arm/Group | A: Letrozole | B,C+D Palbociclib +Letrozole Regimen
Number analyzed (Participants) | 65 | 129
score on a scale | 3.7 (2.3) | 3.6 (2.3)

5. Secondary Outcome: Number and Severity of Adverse Events
Description: To evaluate the overall safety and tolerability for the combination of letrozole and palbociclib. The number of patients experiencing at least one adverse event. Refer to Adverse Events section for more details.
Time Frame: Baseline and weekly through 12 months after randomization
Population: Patients treated with letrozole with palbociclib, i.e. groups B+C+D, were pooled and compared to those treated with letrozole alone (group A). The pooling of groups B-D was pre-planned and defined in the Statistical Analysis Plan.
Measure: Count of Participants; unit: Participants
Groups:
- B+D+C Palbociclib + Letrozole Regimen: Comparison between Group A and Group (B,C+D).
Arm/Group | A: Letrozole | B+D+C Palbociclib + Letrozole Regimen
Number analyzed (Participants) | 100 | 201
Participants | 91 | 199

6. Secondary Outcome: Measurement of Ki67 Marker
Description: To compare Ki67 results after 2 weeks and 14 weeks of study therapy. Log fold change in Ki67 from week 2-week 14.
Time Frame: Week 2 and week 14
Population: Data included for 176 patients that had a 2 week sample.
Measure: Median (Inter-Quartile Range); unit: log fold change in Ki67
Arm/Group | A: Letrozole | B: Letrozole Then Letrozole + Palbociclib | C: Palbociclib Then Letrozole + Palbociclib | D: Letrozole + Palbociclib | B+D+C Palbociclib + Letrozole Regimen
Number analyzed (Participants) | 61 | 39 | 44 | 32 | 115
log fold change in Ki67 | -0.1 [-1.1 to 0.4] | -2.1 [-3.5 to -1.3] | -0.4 [-2.1 to 0.0] | 0.0 [-0.1 to 0.9] | -1.0 [-2.2 to 0.0]

7. Secondary Outcome: Comparison of Surgical Intent (Mastectomy; Breast Conservation)
Description: To compare changes between surgical intent at baseline; surgical intent after 14 weeks; and actual surgery received after treatment with letrozole with or without palbociclib. Percentage of patients change to receiving breast conservation and receiving breast conservation.
Time Frame: Time frame between baseline and surgery date. (Note-surgical intent happened before randomization).
Population: Data included for 268 patients where surgical type and intent was available. Patients treated with letrozole with palbociclib, i.e. groups B+C+D, were pooled and compared to those treated with letrozole alone (group A). The pooling of groups B-D was pre-planned and defined in the Statistical Analysis Plan.
Measure: Count of Participants; unit: Participants
Groups:
- B+D+C Palbociclib + Letrozole Regimen: Comparison between Group A and Groups (B,C+D).
Arm/Group | A: Letrozole | B+D+C Palbociclib + Letrozole Regimen
Number analyzed (Participants) | 90 | 178
Participants
  Change to breast conservation (actual surgery received) from mastectomy (intended at baseline) | 16 | 25
  Breast conservation received (actual surgery) unchanged from what was intended at baseline | 63 | 123
  Change to planned breast conservation (intended at the end of tx) from planned mastectomy | 14 | 25
  Breast conservation planned (at the end of tx) unchanged from what was intended at baseline | 62 | 118

ADVERSE EVENTS:
Time Frame: Baseline and weekly through 12 months after randomization
Description: To evaluate the overall safety and tolerability for the combination of letrozole and palbociclib. Patients treated with letrozole with palbociclib, i.e. groups B+C+D, were pooled and compared to those treated with letrozole alone (group A). The pooling of groups B-D was pre-planned and defined in the Statistical Analysis Plan.
Arm/Group | A: Letrozole | B+D+C Palbociclib + Letrozole Regimen
All-Cause Mortality (participants affected / at risk) | 1/100 | 3/201
Serious Adverse Events (participants affected / at risk) | 3/100 | 17/201
Other Adverse Events (participants affected / at risk) | 91/100 | 199/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Letrozole (N=100) | B+D+C Palbociclib + Letrozole Regimen (N=201)
Cardiac failure (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: Letrozole (N=100) | B+D+C Palbociclib + Letrozole Regimen (N=201)
Anaemia (Blood and lymphatic system disorders) | 3 | 20
Constipation (Gastrointestinal disorders) | 10 | 26
Diarrhoea (Gastrointestinal disorders) | 14 | 33
Dyspepsia (Gastrointestinal disorders) | 7 | 19
Nausea (Gastrointestinal disorders) | 18 | 50
Oral pain (Gastrointestinal disorders) | 1 | 12
Stomatitis (Gastrointestinal disorders) | 0 | 20
Vomiting (Gastrointestinal disorders) | 4 | 14
Fatigue (General disorders) | 41 | 117
Upper respiratory tract infection (Infections and infestations) | 7 | 17
Urinary tract infection (Infections and infestations) | 5 | 15
Contusion (Injury, poisoning and procedural complications) | 7 | 9
Procedural pain (Injury, poisoning and procedural complications) | 5 | 9
Alanine aminotransferase increased (Investigations) | 7 | 23
Aspartate aminotransferase increased (Investigations) | 3 | 15
Blood alkaline phosphatase increased (Investigations) | 6 | 7
Blood creatinine increased (Investigations) | 0 | 10
Neutrophil count decreased (Investigations) | 2 | 110
Platelet count decreased (Investigations) | 0 | 31
White blood cell count decreased (Investigations) | 1 | 49
Decreased appetite (Metabolism and nutrition disorders) | 4 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 9
Dizziness (Nervous system disorders) | 8 | 24
Headache (Nervous system disorders) | 21 | 38
Depression (Psychiatric disorders) | 10 | 9
Insomnia (Psychiatric disorders) | 7 | 16
Breast pain (Reproductive system and breast disorders) | 12 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 26
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 17
Rash (Skin and subcutaneous tissue disorders) | 2 | 12
Hot flush (Vascular disorders) | 40 | 54
Hypertension (Vascular disorders) | 11 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT02296801/Prot_SAP_000.pdf